CLINICAL TRIAL: NCT06163729
Title: A Single-arm, Multicenter Phase II Clinical Study of Camrelizumab Combined With Chemotherapy Followed by Radiotherapy in the Perioperative Treatment of Gastroesophageal Junction Adenocarcinoma
Brief Title: Camrelizumab Combined With Chemotherapy and Radiotherapy Perioperative Treatment of Esophageal Gastric Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shugeng Gao, Vice president, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-OBU-BJ-GC-II-009
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-12

CONDITIONS: Gastroesophageal Junction Adenocarcinoma (Siewert II-III)
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+Oxaliplatin+Paclitaxel (Albumin Bound) +radiotherapy (Experimental)
  Interventions: Drug: Camrelizumab+Oxaliplatin+Paclitaxel (Albumin Bound) +radiotherapy

INTERVENTIONS:
Drug: Camrelizumab+Oxaliplatin+Paclitaxel (Albumin Bound) +radiotherapy — Durg：Camrelizumab: 200mg, iv, d1, q3w Durg ：Oxaliplatin, 100mg/m2 , iv, d1, q3w Durg ：Paclitaxel(Albumin Bound), 125mg/m2, iv, d1, d8, q3w； Durg ：Radiotherapy, PGTV：45.1Gy/2.05Gy/ 22f； PTV：40.04Gy/1.82Gy/ 22f；Five days a week for more than four weeks

SUMMARY:
This project intends to study the efficacy and safety of camrelizumab combined with chemotherapy followed by radiotherapy in the perioperative treatment of AEG.

DETAILED DESCRIPTION:
The incidence of Adenocarcinoma of esophagogastric junction (AEG) is increasing in recent years. According to the statistics of The National Cancer Center of Japan, the proportion of AEG in gastric adenocarcinoma increased from 2.3% in the middle of the 20th century to 10.3% in the beginning of this century, and the proportion of Siewert II in AEG increased from 28.5% to 57.3%. Due to the special biological characteristics of tumor in this region, its definition and surgical treatment principles are controversial.

For AEG, the clinical study results of neoadjuvant chemoradiotherapy + surgery + chemotherapy showed that the tumor stage could be reduced, R0 resection could be improved and overall survival could be improved, without increasing postoperative complications and mortality. Long-term follow-up results from the German TRIAL III of preoperative chemoradiotherapy for AEG (POET) showed that preoperative chemoradiotherapy reduced recurrence (5y-local recurrence: 21% vs. 38%) and prolonged survival (3y-OS: 46.7% vs. 26.1%), without a significant increase in treatment toxicity and perioperative complications . Although some patients with AEG were included in the resolve 、 prodigy and resolution study ,and the total population could benefit from postoperative adjuvant radiotherapy and chemotherapy, but it was uncertain whether the patients with AEG could benefit in Asia.

Therefore, this project intends to study the efficacy and safety of camrelizumab combined with chemotherapy followed by radiotherapy in the perioperative treatment of AEG.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged from 18 to 80 years old;
2. Patients with pathologically confirmed gastroesophageal junction adenocarcinoma (Siewert II-III)
3. Resectable tumors with staging t3-4N0M0 or T1-4N+M0 confirmed by CT or MRI according to AJCC version 8 staging System;
4. Disease must be measurable by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1);
5. No prior anti-tumor therapy, including surgery, chemotherapy, radiotherapy, targeted and immunotherapy;
6. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1 at trial entry;
7. Estimated life expectancy of more than 3 months;
8. Adequate haematological, hepatic and renal functions defined by the protocol;
9. Prior use of anti-tumor traditional Chinese medicine, proprietary Chinese medicine, immunomodulators (such as thymosin, interleukin, etc.) must be ≥2 weeks from the beginning of the study
10. Negative blood pregnancy test at Screening for women of childbearing potential; Highly effective contraception for both male and female subjects if the risk of conception exists;
11. The subjects participated in the study voluntarily, fully understood and informed the study and signed the informed consent;

Exclusion Criteria:

1. Previous malignant disease within the last 5 years with the exception of basal or squamous cell carcinoma of the skin or carcinoma in situ (bladder, cervical, colorectal, breast)；
2. Any active autoimmune disease or history of autoimmune disease (such as interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (can be included after hormone replacement therapy)); The subjects with childhood asthma who had been completely relieved and did not need any intervention or vitiligo in adulthood could be included, but the subjects who needed bronchodilator for medical intervention could not be included;
3. Patients with congenital or acquired immune deficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV DNA ≥ 500 IU / ml), hepatitis C (HCV antibody positive and HCV-RNA higher than the detection limit of the analytical method), or co infection of hepatitis B and hepatitis C;
4. Active tuberculosis;
5. Prior organ transplantation, including allogeneic stem-cell transplantation；
6. Other protocol-defined inclusion/exclusion criteria could apply.
7. Used immunosuppressive drugs within 14 days before the first dose of study drug, excluding nasal and inhaled corticosteroids or physiological doses of systemic corticosteroids;
8. Accination with live or live/attenuated viruses within 4 weeks of the first dose of camrelizumab and while on trial is prohibited except for administration of inactivated vaccines;
9. History of uncontrolled intercurrent illness including hypertension, active infection, diabetes , hereditary bleeding , coagulopathy with a risk of bleedingor, cardiac diseases or symptoms;
10. Patients with past and current interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-associated pneumonia, and severe impaired lung function may interfere with the detection and management of suspected drug-associated pulmonary toxicity;
11. Known history of allergy to the drug components of this regimen;
12. Presence of unresectable factors, including tumor, contraindications to surgery, or rejection of surgery;
13. Major surgical procedures were performed within 4 weeks prior to initial administration;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (PCR) | 4 weeks after surgery
  pCR rate is defined as the percentage of patients, relative to the total of enrolled subjects,achieving complete histological regression with no available tumor cells yT0N

SECONDARY OUTCOMES:
3 years-Overall Survival (3y-OS) | up to 3 years
  Percentage of patients who survived 3 years after the start of randomized treatment
years-Event free survival (3y-EFS) | up to 3 years
  Proportion of patients with event-free survival at 3 years after randomization
Disesease free survival（DFS） | up to 3 years
  Proportion of patients with disease-free survival at 3 years after randomization
Number of Subjects With Treatment-Emergent Adverse Events (TEAEs) According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 | From the the first dose of study drug administration up to 28 days after the last dose of study drug administration, assessed up to 1 years
  TEAEs will be defined as the adverse events (AEs) that occur between first dose of study drug administration and 28 days after the last dose of study drug administration that were absent before treatment or that worsened relative to pretreatment state.
R0 resection rate | 24 months
  R0 resection rate is defined as the percentage of patients, relative to the total of enrolled subjects, undergoing R0 resection of primary tumour

CONTACTS AND LOCATIONS:
Locations (1):
- Shugeng Gao, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No